CLINICAL TRIAL: NCT06294340
Title: Noise, Oxidative Stress and Cardiovascular System
Acronym: NOXYCARD
Status: Not yet recruiting | Type: Observational
Sponsor: University of Belgrade (Other)
Responsible Party: Principal Investigator, Katarina Paunovic, Professor, University of Belgrade
Other Study IDs: 1322-IX/42
Record Dates: First submitted 2024-02-19; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Noise; Adverse Effect; Noise Exposure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with normal body weight: The effects of noise exposure on blood pressure, cardiovascular and hemodynamic parameters, stress hormones, and markers of oxidative stress and inflammation in individuals with normal body weight.
  Interventions: Other: Exposure to loud pre-recorded road traffic noise
- Overweight / obese participants: The effects of noise exposure on blood pressure, cardiovascular and hemodynamic parameters, stress hormones, and markers of oxidative stress and inflammation in individuals with overweight/obesity.
  Interventions: Other: Exposure to loud pre-recorded road traffic noise

INTERVENTIONS:
Other: Exposure to loud pre-recorded road traffic noise — Participants of both arms will be exposed to the same loud pre-recorded road traffic noise in a laboratory setting.

SUMMARY:
Environmental noise represents a health problem for at least one in five citizens of the European Union. Noise exposure leads to the development of arterial hypertension, myocardial infarction, stroke, and obesity. Given the limited information on noise exposure and noise effects on humans in the Republic of Serbia, the overall objective of NOXYCARD is to collect environmental noise levels data; to identify long-term and short-term noise effects on the cardiovascular system; and to evaluate the levels of blood stress hormones, oxidative stress, and inflammation in individuals with normal body weight and individuals with obesity.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65
* both genders
* good self-reported health

Exclusion Criteria:

* diabetes mellitus
* arterial hypertension or other cardiovascular diseases
* kidney diseases
* pregnancy
* malignant diseases
* mental diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All persons who visit the Nutrition Counselling Unit of the Institute of Hygiene and Medical Ecology, located at the Faculty of Medicine, University of Belgrade will be eligible to participate in the study. The study population will include 75 participants with normal weight and 75 overweight/obese participants who meet the inclusion criteria for the survey. Participants will be informed of the protocol and sign an informed consent form.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Systolic blood pressure | 10, 40, and 50 minutes
  Systolic blood pressure in mmHg, higher values indicate high risk
Concentration of stress hormone | 10, 40, and 50 minutes
  Cortisol level in mcg/dL, higher values indicate high risk

SECONDARY OUTCOMES:
Diastolic blood pressure | 10, 40, and 50 minutes
  Diastolic blood pressure in mmHg, higher values indicate high risk
Concentration of inflammation parameters | 10, 40, and 50 minutes
  Interleukin-1-Beta levels in pg/mL, higher values indicate high risk

CONTACTS AND LOCATIONS:
Overall Officials: Katarina Paunovic, MD, PhD, Principal Investigator — University of Belgrade
Locations (1):
- Faculty of Medicine, University of Belgrade, Belgrade, Beograd, Serbia

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared. Data will be shared in cumulative form.

REFERENCES:
- [Result] Paunovic K, Jakovljevic B, Stojanov V. The timeline of blood pressure changes and hemodynamic responses during an experimental noise exposure. Environ Res. 2018 May;163:249-262. doi: 10.1016/j.envres.2018.01.048. Epub 2018 Feb 22. PMID 29459307
- [Result] Paunovic K, Stojanov V, Jakovljevic B, Belojevic G. Thoracic bioelectrical impedance assessment of the hemodynamic reactions to recorded road-traffic noise in young adults. Environ Res. 2014 Feb;129:52-8. doi: 10.1016/j.envres.2014.01.001. Epub 2014 Jan 25. PMID 24529003